CLINICAL TRIAL: NCT02530255
Title: Evaluation of an Oral Telomerase Activator on Retinal Amyloid
Brief Title: Telomerase Activator and Retinal Amyloid
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chippewa Valley Eye Clinic (Other)
Collaborators: TA-Sciences (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TAS-003-AD
Record Dates: First submitted 2015-07-25; First posted 2015-08-21 (Estimated); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Alzheimer Disease
Keywords: retinal amyloid; Retinal amyloid index; Alzheimer disease; telomere attrition; telomere activation
MeSH Terms: conditions — Alzheimer Disease | interventions — cycloastragenol; Cellulose

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Study subjects receiving placebo: Intervention - two capsules, one morning and one night for one year; placebo for cycloastragenol
  Interventions: Dietary Supplement: placebo (for cycloastragenol)
- cycloastragenol (Active Comparator): Study subjects receiving cycloastragenol: Intervention - cycloastragenol; oral capsules 8mg. per day (two capsules) one in the morning and one at night for one year.
  Interventions: Dietary Supplement: cycloastragenol

INTERVENTIONS:
Dietary Supplement: cycloastragenol — Oral telomerase activator - cycloastragenol.
  Other Names: TA-65
  Arms: cycloastragenol
Dietary Supplement: placebo (for cycloastragenol) — placebo comparator, placebo for cycloastragenol.
  Other Names: Silicone dioxide and cellulose
  Arms: Placebo

SUMMARY:
A method of detecting amyloid in the retina has been developed. A specially designed retinal camera will directly visualze and record retinal amyloid and via image processing will generate a number: the retinal amyloid index (RAI). The amount of retinal amyloid correlates with cerebral amyloid and has a predictive value in Alzheimer's disease.

Telomere attrition accounts for cellular aging and is felt to have a pivotal role in Alzheimer's disease. The investigators plan to screen individuals to select those having retinal amyloid then evaluate an oral telomerase activator to determine if its use can alter the RAI over time compared to placebo.

DETAILED DESCRIPTION:
Telomerase Activation - Retinal Amyloid Study

Telomere attrition has been linked to the neurodegenerative disease Alzheimer's disease (AD). AD is definitively diagnosed at autopsy a fact that has prompted exhaustive investigations looking for reliable biomarkers of AD. It is known that the clinical signs of AD are the end result of years of accumulation of an aggregated protein substance, amyloid. The retina is part of the brain and recently, a diagnostic technology has been developed that allows detection of retinal amyloid. Tissue studies show a correlation between retinal and cerebral amyloid, and it has been proposed that early detection of retinal amyloid, long before clinical dementia, may offer an opportunity for intervention to slow or halt progressive amyloid deposition. Special imaging technology has been developed that is capable of detecting retinal amyloid via an adapted retinal camera. Neurovision Imaging (NVI) is the company that has developed these testing technologies: both for retinal amyloid detection and measurement.

A study is proposed that will investigate if there is a measurable treatment effect of the telomerase activator TA-65 on retinal amyloid of the participants. It is anticipated that recruiting will primarily be directed at adult children of individuals with clinical AD.

The study will include 50 participants and will have a term of 12 months; it is anticipated that up to 300 individuals will be screened to acquire the participants. The study will be conducted at a single site: Chippewa Valley Eye Clinic, Eau Claire, Wisconsin and/or its satellites. TA-Sciences will sponsor the study, provide telomere length testing on saliva samples collected at the start and conclusion of study. TA-Sciences will also provide active and placebo product for term of study.

ELIGIBILITY:
Inclusion Criteria:

* qualifying retinal amyloid index (RAI) number as determined at screening
* Must be able to swallow capsule

Exclusion Criteria:

* Cancer treatment within 5 years (except non-melanoma skin cancer)
* Must be able to swallow capsule

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Retinal Amyloid Index (RAI) | one year.
  Measurement of amyloid fluorescence while taking cycloastragalone or placebo

SECONDARY OUTCOMES:
Telomere length (kilobases) | one year
  Telomere length measured in white blood cells isolated from saliva

CONTACTS AND LOCATIONS:
Overall Officials: Coad T. Dow, M.D., Principal Investigator — Chippewa Valley Eye Clinic
Locations (1):
- Chippewa Valley Eye Clinic, Eau Claire, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Boccardi V, Pelini L, Ercolani S, Ruggiero C, Mecocci P. From cellular senescence to Alzheimer's disease: The role of telomere shortening. Ageing Res Rev. 2015 Jul;22:1-8. doi: 10.1016/j.arr.2015.04.003. Epub 2015 Apr 17. PMID 25896211
- [Background] Koronyo Y, Salumbides BC, Black KL, Koronyo-Hamaoui M. Alzheimer's disease in the retina: imaging retinal abeta plaques for early diagnosis and therapy assessment. Neurodegener Dis. 2012;10(1-4):285-93. doi: 10.1159/000335154. Epub 2012 Feb 10. PMID 22343730
- [Background] Mattson MP. Emerging neuroprotective strategies for Alzheimer's disease: dietary restriction, telomerase activation, and stem cell therapy. Exp Gerontol. 2000 Jul;35(4):489-502. doi: 10.1016/s0531-5565(00)00115-7. PMID 10959037
- [Background] Panossian LA, Porter VR, Valenzuela HF, Zhu X, Reback E, Masterman D, Cummings JL, Effros RB. Telomere shortening in T cells correlates with Alzheimer's disease status. Neurobiol Aging. 2003 Jan-Feb;24(1):77-84. doi: 10.1016/s0197-4580(02)00043-x. PMID 12493553
- [Background] Wang J, Zhao C, Zhao A, Li M, Ren J, Qu X. New insights in amyloid beta interactions with human telomerase. J Am Chem Soc. 2015 Jan 28;137(3):1213-9. doi: 10.1021/ja511030s. Epub 2015 Jan 17. PMID 25564872